CLINICAL TRIAL: NCT00451945
Title: New Indications for Ultrasound in the Staging of Cervical Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-KF 2007-004
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Biopsy; Ultrasonography; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: biopsy
Device: 3d-ultrasound and fusion of UL and PET/CT

SUMMARY:
The purpose is to investigate and evaluate two new diagnostic methods using ultrasound in the staging of cervical cancer.

1. 3-D-ultrasound of the tumour to estimate its volume and local spread
2. Fusion of PET/CT and ultrasound to evaluate and biopsy lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer,
* PET/CT pos. lymph nodes,
* Patients over 18 years old

Exclusion Criteria:

* Pregnancy,
* Lactating,
* Diabetic

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2007-03; Study Completion 2008-03

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Nielsen, MDSc, Principal Investigator — Department of radiology, section of ultrasound
Locations (1):
- Copenhagen univercity hospital, Department of Radiology, section of ultrasound, Copenhagen, Denmark